CLINICAL TRIAL: NCT03311568
Title: Microcirculatory Alterations in Critical Disease. New Ultrasound Technology for Assessment of Small-vessel Circulation Pathophysiology
Brief Title: Microcirculatory Alterations in Critical Disease: New Ultrasound Technology
Acronym: SepCease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Researcher has quit. Question still unanswered. A related study (observational, not to be registered) has started recently.
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017/908
Record Dates: First submitted 2017-10-11; First posted 2017-10-17 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Critical Illness; Septic Shock
Keywords: Ultrasonography; Microvessels; Physiopathology; Diagnostic Imaging; Critical Care
MeSH Terms: conditions — Critical Illness; Shock, Septic | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Prospective observational study. Validation of a new non-invasive ultrasound device in four controlled categories of study participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- surgery in general anaesthesia (Experimental): 10 patients. ultrasound for microcirculatory assessment applied.
  Interventions: Device: ultrasound for microcirculatory assessment
- open chest cardiac surgery (Experimental): 10 patients. ultrasound for microcirculatory assessment applied.
  Interventions: Device: ultrasound for microcirculatory assessment
- critical septic shock at ICU (Experimental): 20 patients. ultrasound for microcirculatory assessment applied.
  Interventions: Device: ultrasound for microcirculatory assessment
- healthy volunteers (Experimental): 10 subjects. ultrasound for microcirculatory assessment applied.
  Interventions: Device: ultrasound for microcirculatory assessment

INTERVENTIONS:
Device: ultrasound for microcirculatory assessment — Ultrasound for microcirculatory assessment Repeated measurements within study participants for analysis of variance and explorative analyses of ultrasound signals, to identify most suitable parameters to describe microcirculatory alterations in critical disease, especially in sepsis.
  Analyse blood flow velocities in several depths and from several vessels of different sizes simultaneously
  US registration repeated within each study participant consecutively on seven different regions of the body surface.

SUMMARY:
Aim of this study is (1) to test and further develop a new non-invasive ultrasound method, and (2) to gain new insight into microcirculatory alterations during critical disease, particularly in critical septic shock patients.

Although early identification and treatment of sepsis have had top priority among the working tasks of the international 'Surviving Sepsis Campaign' society (collaboration of the Society of Critical Care Medicine and the European Society of Intensive Care Medicine) for several years, which have led to improved survival over the last two decades, there is no objective validated diagnostic test to identify or to support the clinical diagnosis at an early stage. Analogous, there is no validated monitoring system available to guide and evaluate the effects of stabilizing measurements in sepsis, or other critical disease, at the microcirculatory level. And thus, there is an enormous knowledge gap regarding dynamic changes at the microcirculatory level during sepsis and other critical disease.

Goal with this study is to investigate the robustness of this new US-technology, regarding its ability to identify and monitor critical microcirculatory impairment during critical disease. The investigators believe this technology may improve early diagnosis and thus early initiation of adequate treatment in septic shock. Its mobile and non-invasive qualities, as in most ultrasound methods, substantiate its availability to a wide range of clinical settings.

DETAILED DESCRIPTION:
Critical disease, e.g. life threatening septic shock triggered from infections with multiorgan failure, demands aggressive medical treatment in specialized intensive care units (ICU). Incidences and mortality of sepsis vary significant, depending on regional medical culture, diagnostic criteria and the time span and method of data collection.

Common clinical appearance of critical disease is often life threatening low blood pressure, impaired consciousness up to coma, abnormal breathing patterns, and then subsequently secondary organ failures which further increases mortality. The influence of these 'macro-haemodynamic symptoms', i.e. physiologic aberrations that can be assessed using standard patient monitoring systems, on the tissue micro-circulation where organ damage and finally cell death occurs, is only indirectly available for assessment. Basically, the coarse therapeutic approach to circulatory shock is to normalize macro-haemodynamic parameters, without any robust method to evaluate and monitor micro-circulatory effects. Thus, following current guidelines and clinical practice, it is sometimes not known for sure, on an individual basis, whether treatment and stabilization measures increase survival chances.

Studies of the microcirculation have been performed using invasive micro-dialysis, direct orthogonal polarization spectral imaging and direct side-stream dark-field microscopy. The wide use of these methods is challenged by the fact that they are very expensive and demand extended operator expertise.

The investigators think there is sufficient evidence to claim that further improvement in early diagnostic and therapy guidance of sepsis, septic shock and other critical disease, depends on increased knowledge of microcirculatory alterations, and widespread affordable technical solutions to detect and monitor the course of sepsis and other critical disease at the microcirculatory level.

At the Norwegian University of Technology and Science (NTNU), Department of Circulation and Medical Imaging (ISB), new ultrasound technology has been developed by Professor Hans Torp, which may offer an operator-independent, affordable and non-invasive method to evaluate microcirculation in humans.

In general, ultrasound is unique in that sense that it facilitates non-invasive imaging of anatomy and physiology. The unique with this new probe is the emittance of ultrasound waves from the whole cross-section of the probe surface.

To describe the expected spectrum of microcirculatory impairment during different stages of sepsis, septic shock and comparable critical disease, firstly US registrations are needed from persons with known normal microcirculation. Then, registrations of normal microcirculation are needed in persons exposed to increasing amounts of circulatory stress. Finally, microcirculatory conditions will be observed in patients with critical septic shock. Thus, firstly healthy volunteers are included, then stabile patients undergoing major planned surgery, and finally patients in critical septic shock demanding advanced intensive care treatment and monitoring.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers: No disease, no medication, no history of cardiovascular events, no smoking, body mass index (BMI) 20-35 kg/m2, no premature cardiovascular disease among parents.
* patients scheduled for non-thoracic surgery in general anesthesia: BMI 20-35 kg/m2, surgery scheduled for general anaesthesia/narcosis without any expected complications. Typical candidates: Laparotomy/laparoscopy. Cholecystectomy, adnexectomy, hysterectomy. No disease other than the indication for surgery, no medication other than those needed for the present condition demanding surgery, e.g. antibiotics, pain medicine.
* scheduled for open-chest cardiac surgery, Age < 60 years, BMI 20-35 kg/m2, no diagnosed peripheral artery disease, no history of cardiovascular events other than those indicating the actual surgery - 'as healthy as possible', meaning no previous cardiac surgery, no cerebral vascular events, no diagnosed peripheral artery disease. These patients mostly have a history of hypertension, diabetes, hypercholesterolaemia, myocardial infarction or at least angina pectoris, as well as the associated medical therapy. Typical candidates: Coronary artery disease patients without other diagnosed vascular disease.
* septic shock defined as 1) suspected infection, and 2) an acute change in the 'Sequential (Sepsis-Related) Organ Failure Assessment' score (SOFA) of two or more points and serum-lactate acid above 2mmol/l and 3) at least one vasopressor (strong blood-pressure stimulating medical infusion) required to maintain mean blood pressure (MAP) above 65 mmHg, despite adequate fluid resuscitation. Mechanical ventilation ('Respirator'). Advanced invasive haemodynamic monitoring including continuous invasive arterial blood pressure, central venous pressure, pulmonary artery pressure (pulmonary artery catheter/ 'Swan Ganz'), cardiac output and systemic vascular resistance monitoring, as well as circulatory parameters associated with these monitoring systems. Frequent non-invasive cardiac ultrasound - echocardiography ('Echo'). Typical candidates: Critical disease ICU patients with suspected septic shock.

Exclusion Criteria:

* Healthy volunteers: Pregnancy, age > 40 years or < 20 years, BMI < 20 or BMI > 35, history of cardiovascular disease, diabetes or hypertension or previous/ongoing pharmacological/non-pharmacological therapy for such diseases. Hereditary vascular disease or connective tissue disease. Skin disease suspected to be influenced by or to influence US registrations (skin-probe interactions)
* non-thoracic surgery: Pregnancy, age > 40 years, BMI < 20 or BMI > 35, smoking, history of cardiovascular disease/events, diabetes or hypertension or previous/ongoing pharmacological/non-pharmacological therapy for such diseases. Hereditary vascular disease or connective tissue disease. Skin disease suspected to be influenced by or to influence US registrations (skin-probe interactions).
* open-chest cardiac surgery: Pregnancy, age > 60 years, BMI < 20 or BMI > 35, history of open chest cardiac surgery. Hereditary vascular disease or connective tissue disease.
* septic shock: Pregnancy. History of heart failure and ongoing medical therapy for such disease. Hereditary vascular disease or connective tissue disease. Palliative or proliferated cancer disease. Advanced skin disease complicating performance of the US registrations. Isolated contagious patients and patients isolated due to a pronounced immune-suppressed state of health.
* General: study equipment or ultrasound registrations are suspected to disturb patient treatment
* General: consent refused by patient or (in case of septic shock) by family member next to kin

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Pulsatile index | 1 day
  (velocity max - velocity min) / mean velocity
Time-velocity-integral | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Hans Torp, prof, Study Chair — Norwegian University of Science and Technology; Daniel Bergum, md phd, Principal Investigator — St. Olavs Hospital
Locations (1):
- St Olavs Hospital, Dept Gastrointestinal Surgery, Dept Thoracic Surgery, Dept Intensive Care Medicine, Trondheim, Norway